CLINICAL TRIAL: NCT04058275
Title: "Immunomodulation in GWI (Phlebotomy)"
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Georgetown University (Other)
Collaborators: Nova Southeastern University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-0470
Record Dates: First submitted 2019-08-02; First posted 2019-08-15 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Gulf War Illness
MeSH Terms: interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Deployed to 1990-1991 Persian Gulf War Do not meet Kansas Criteria for Gulf War Illness [Steele L. Prevalence and patterns of Gulf War illness in Kansas veterans: association of symptoms with characteristics of person, place, and time of military service. Am J Epidemiol. 2000 Nov 15; 152:992-1002. PubMed PMID: 11092441.] Good general medical and psychiatric health
  Interventions: Other: Draw blood (phlebotomy, 83 ml)
- Gulf War Illness: Deployed to 1990-1991 Persian Gulf War Meet Kansas Criteria for Gulf War Illness [Steele L. Prevalence and patterns of Gulf War illness in Kansas veterans: association of symptoms with characteristics of person, place, and time of military service. Am J Epidemiol. 2000 Nov 15; 152:992-1002. PubMed PMID: 11092441.] plus Center for Disease Control criteria for Chronic Multisymptom Illness (CMI) [Fukuda K, Nisenbaum R, Stewart G, Thompson WW, Robin L, Washko RM, Noah DL, Barrett DH, Randall B, Herwaldt BL, Mawle AC, Reeves WC. Chronic multisymptom illness affecting Air Force veterans of the Gulf War. JAMA. 1998 Sep 16;280(11):981-8. PubMed PMID: 9749480.]
  Interventions: Other: Draw blood (phlebotomy, 83 ml)

INTERVENTIONS:
Other: Draw blood (phlebotomy, 83 ml) — Draw 83 ml of blood
  Other Names: phlebotomy

SUMMARY:
Gulf War Illness and deployed veterans of the 1990-1991 Persian Gulf War are invited to have a brief history and physical examination to determine their health status, complete questionnaires, then donate about 83 ml of blood. There is no follow-up

DETAILED DESCRIPTION:
Gulf War Illness and deployed veterans of the 1990-1991 Persian Gulf War are invited to have a brief history and physical examination to determine their health status, complete questionnaires, then donate about 83 ml of blood. There is no follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Kansas Criteria for GWI
* CDC criteria for CMI

Exclusion Criteria:

* Chronic medical or psychiatric disorder that may be responsible for symptoms of GWI

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Deployed veterans
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Gene expression in peripheral blood mononuclear cells | After study recruitment, phleobotomy and mRNA quantification for all participants has been completed in June 2020
  Determine mRNA expression in peripheral blood mononuclear cells (PBMCs)

CONTACTS AND LOCATIONS:
Overall Officials: James N Baraniuk, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided
Cell counts and mRNA levels in peripheral blood mononuclear cells will be available for analysis by contacting the PI